CLINICAL TRIAL: NCT07233720
Title: A Multicenter Prospective Real-world Study of Zanubrutinib Combined With Rituximab (ZR) in the First-line Treatment for Patients With Marginal Zone Lymphoma (MZL)
Brief Title: Zanubrutinib Combined With Rituximab in the Treatment for Patients With Marginal Zone Lymphoma
Status: Recruiting | Type: Observational
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Zhihua Yao, PhD, Director, Henan Cancer Hospital
Other Study IDs: HNSZLYYNHL10
Record Dates: First submitted 2025-07-08; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-10

CONDITIONS: Marginal Zone Lymphoma
Keywords: Marginal Zone Lymphoma; Zanubrutinib; Rituximab
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone | interventions — zanubrutinib; Rituximab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Zanubrutinib Combined With Rituximab: Induction treatment:
  Rituximab, 375mg/m2, Intravenous administration on day 1 (21 days/cycle); Zanubrutinib, 160mg twice daily continuous oral administration from 1 to 8 cycles (21 days/cycle)
  Maintenance treatment:
  Zanubrutinib, 160mg twice daily continuous oral administration for two years (28 days/cycle)
  Interventions: Drug: Zanubrutinib; Drug: Rituximab

INTERVENTIONS:
Drug: Zanubrutinib — 160mg twice daily continuous oral administration.
  Other Names: Zanubrutinib pills
Drug: Rituximab — 375mg/m2, Intravenous administration on day 1 of each 3-week cycle
  Other Names: RiTUXimab Injection

SUMMARY:
This is a prospective single arm, multi-center, real-world study to observe the efficacy and safety of ZR (Zanubrutinib combined with Rituximab) in the first-line treatment for patients with marginal zone lymphoma (MZL).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with CD20-positive marginal zone lymphoma diagnosed by histopathology
2. First-line treatment with the combination regimen of zanubrutinib and rituximab
3. No receiving systematic treatment before enrollment
4. Having at least one measurable lesions. Measurable lesions were defined as: the longest diameter of lymph node lesions in CT cross-sectional images > 1.5 cm, or the longest diameter of the extranodal lesion is greater than 1.0cm
5. The patients voluntarily joined this study, signed the informed consent form, had good compliance and cooperated with the follow-up.

Exclusion Criteria:

1. Other malignant tumor history or active malignant tumor need be treated
2. In addition to zanubrutinib and rituximab, other anti-tumor drug treatments were also received simultaneously (except for glucocorticoids aimed at controlling symptoms before formal treatment).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with CD20-positive marginal zone lymphoma diagnosed by histopathology for first-line treatment.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-11-18 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
complete response rate | every 6 weeks from the day of the first cycle of induction chemotherapy treatment (each cycle is 21 days) and every 8 weeks from the day of the first cycle of maintenance treatment (each cycle is 28 days) to 18 months after last patient's enrollment
  the total proportion of patients with complete response (CR)

SECONDARY OUTCOMES:
objective response rate | every 6 weeks from the day of the first cycle of induction chemotherapy treatment (each cycle is 21 days) and every 8 weeks from the day of the first cycle of maintenance treatment (each cycle is 28 days) to 18 months after last patient's enrollment
  the total proportion of patients with complete response (CR) and partial response (PR)
progression-free survival | from the day of the first cycle of treatment to the date of confirmed progressive disease or death, whichever occurs first after last patient's enrollment (each cycle is 21 days for induction treatment, and 28 days for maintenance treatment)
  the total proportion of patients with no progression from date of the first day of treatment to the date of confirmed progressive disease or death which one occurs first
overall survival | from date of the first cycle of treatment to the date of death from any cause (each cycle is 21 days for induction treatment, and 28 days for maintenance treatment)
  from date of first day of treatment to the date of death by any cause
incidence and relationship with study drugs of grade 3-4 adverse events | from the date of the first cycle of treatment to 24 months after last patient's enrollment (each cycle is 21 days for induction treatment, and 28 days for maintenance treatment)
  the incidence and relationship with study drugs of grade 3 or 4 adverse events (based on NCI CTC-AE v5.0)

CONTACTS AND LOCATIONS:
Overall Officials: Zhihua Yao, M.D. Ph.D, Study Director — Henan Cancer Hospital
Locations (1):
- Henan Cancer Hospital/The affiliated Cancer Hospital of ZhengZhou university, Zhengzhou, Henan, China